CLINICAL TRIAL: NCT07331272
Title: An Open-label Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of LUCAR-G79D in Subjects With Relapsed/Refractory Systemic Lupus Erythematosus (r/r SLE) and Idiopathic Inflammatory Myopathies (r/r IIM)
Brief Title: A Study of LUCAR-G79D in Subjects With Relapsed/Refractory Systemic Lupus Erythematosus (r/r SLE) and Idiopathic Inflammatory Myopathies (r/r IIM)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nanjing Legend Biotech Co. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LB2404D-0001
Record Dates: First submitted 2025-12-15; First posted 2026-01-09 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Systemic Lupus Erythematosus (SLE); Idiopathic Inflammatory Myopathies(IIM)
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Myositis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chimeric antigen receptor T cells (LUCAR-G79D) (Experimental): Each subject will be given a single-dose LUCAR-G79D cells infusion at each dose level.
  Interventions: Biological: LUCAR-G79D T cells

INTERVENTIONS:
Biological: LUCAR-G79D T cells — Prior to infusion of the LUCAR-G79D T cells, subjects will receive a conditioning premedication regimen consisting of cyclophosphamide and fludarabine.

SUMMARY:
This is a prospective, single-arm, open-label and dose-escalation investigator initialed study to evaluate LUCAR-G79D in adult subjects with r/r SLE and r/r IIM.

DETAILED DESCRIPTION:
This is a prospective, single-arm, open-label clinical study to evaluate the safety, tolerability, pharmacokinetics and efficacy profiles of LUCAR-G79D, a chimeric antigen receptor (CAR) -T cell therapy in subjects with r/r SLE and r/r IIM. Patients who meet the eligibility criteria will receive LUCAR-G79D infusion. The study will include the following sequential stages: screening, pre-treatment (lymphodepleting chemotherapy), treatment (LUCAR-G79D infusion) and follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntary agreement to provide written informed consent.
2. Aged 18 to 70 years, either sex.
3. Adequate organ function meet screening criteria.
4. Positive test for cluster of differentiation antigen 19 (CD19).

SLE:

* Have been diagnosed of SLE at least 6 months before screening.
* At screening, antinuclear antibody, and/or anti-dsDNA antibody, and/or anti-Smith antibody should be positive.
* Fulfill relapsed/refractory SLE conditions.

IIM:

* Have been diagnosed of IIM before screening.
* Positive test for myositis-associated antibodies or myositis-specific antibodies at screening.
* Fulfill relapsed/refractory IIM conditions.

Exclusion Criteria:

1. Active infections such as hepatitis and tuberculosis.
2. Other autoimmune diseases.
3. Serious underlying diseases such as tumor, uncontrolled diabetes.
4. Female subjects who were pregnant, breastfeeding.
5. Those with a history of major organ transplantation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2026-01-29 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence, severity, and type of treatment-emergent adverse events (TEAEs) | 2 years after LUCAR-G79D infusion (Day 1)
Incidence of dose-limiting toxicity (DLT) | 2 years after LUCAR-G79D infusion (Day 1)
Maximum concentration (Cmax) in peripheral blood | 2 years after LUCAR-G79D infusion (Day 1)
Time of maximum concentration (Tmax) in peripheral blood | 2 years after LUCAR-G79D infusion (Day 1)
Area under the concentration-time curve (AUC) in peripheral blood | 2 years after LUCAR-G79D infusion (Day 1)
Recommended Dose regimen finding | 2 years after LUCAR-G79D infusion (Day 1)

SECONDARY OUTCOMES:
Change in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) scores from baseline up to 52 weeks for r/r SLE subjects | 52 weeks after LUCAR-G79D infusion (Day 1)
  SLEDAI-2K is a scale ranging from 0 to 105 points, with higher scores indicating stronger disease activity
Change in manual muscle testing (MMT-8) scores from baseline up to 52 weeks for r/r IIM subjects | 52 weeks after LUCAR-G79D infusion (Day 1)
  MMT-8 is a scale ranging from 0 to 80 points, with higher scores indicating greater preserved muscle strength
Changes from baseline in peripheral blood immunoglobulins from baseline up to 52 weeks for all subjects | 52 weeks after LUCAR-G79D infusion (Day 1)
  Including IgG、IgM、IgA、IgE
Changes from baseline in anti-drug antibody from baseline up to 52 weeks for all subjects | 52 weeks after LUCAR-G79D infusion (Day 1)

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - The Third The People's Hospital of Bengbu, Bengbu, Anhui
  - Nanfang Hospital, Guangzhou, Guangdong
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi

IPD SHARING:
Plan to Share IPD: No